CLINICAL TRIAL: NCT03635515
Title: Post-operative Pain Following Treatment Using the Gentlewave System
Brief Title: Occurrence of Post-op Pain Following Gentlewave
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DENT-2018-26373
Record Dates: First submitted 2018-08-10; First posted 2018-08-17 (Actual); Results first posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-01

CONDITIONS: Root Canal Infection; Endodontic Disease; Endodontic Inflammation; Post-Operative Pain
MeSH Terms: conditions — Dental Pulp Diseases; Pulpitis; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Patients will be asked to indicate their peak pain level in the twenty-four hours prior to the appointment using a visual analog scale (VAS). The VAS scale will consist of a 100mm line where 0 equals 'no pain' and 100 equals the 'worst pain imaginable'. Patients will be divided into one of two treatment groups, either standard cleaning protocol or Gentlewave irrigation. Patient demographics, anesthesia, cleaning and shaping instruments, irrigation technique, and obturation method and material will be recorded, along with the number of appointments, extent of treatment rendered, and the occurrence of over-instrumentation or overfill of obturation material. Once obturation is completed, patients will be given the same VAS scale to take home and asked to record their level of pain at 6, 24, 72, and 168 hours post-treatment.
Who Masked: Participant
Masking Description: Participants will not know which study arm/intervention group they will be assigned to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard Protocol (Control) Group (Active Comparator): Patients will be given a VAS scale to record their highest level of pain 6 hrs prior to treatment. The standard endodontic protocol will be followed. The same VAS scale from pretreatment will be used to record pain level at 6, 24, 72, and 168 hours post-treatment.
  Interventions: Procedure: Standard Endodontic Protocol
- Gentlewave Treatment Group (Active Comparator): Patients will be given a VAS scale to record their highest level of pain 6 hrs prior to treatment. The standard endodontic protocol will be followed through working length verification. For the Gentlewave treatment group, each canal will be shaped to a canal size of 20.06 and to 0.5 - 1mm short of the apical terminus. An occlusal platform will be prepared using the Kool-dam material recommended by Sonendo. The Gentlewave system will be held on the tooth by the clinician and will cycle through five minutes of 3% sodium hypochlorite, two minutes of 8% EDTA, and a final rinse of distilled water. Canals will be obturated with root canal sealer and gutta-percha. The same VAS scale from pretreatment to take home and asked to record their level of pain at 6, 24, 72, and 168 hours post-treatment.
  Interventions: Device: Gentlewave

INTERVENTIONS:
Device: Gentlewave — The Gentlewave system from Sonendo is a FDA cleared root canal irrigation device that uses broad spectrum acoustic energy, internally degassed distilled water, 3% NaOCl, and 8% EDTA to allow for a more thorough cleaning within the tooth. The fluids work to remove necrotic tissue, debris, biofilm, and bacteria while leaving dentin intact and preserving tooth structure. The Gentlewave irrigation replaces the NaOCl ultrasonic activation and EDTA steps of the standard endodontic protocol. Use of the Gentlewave system is contraindicated in teeth with immature apices, teeth with insufficient coronal structure, and teeth with root apices extending into the maxillary sinus.
  Arms: Gentlewave Treatment Group
Procedure: Standard Endodontic Protocol — The tooth will be sufficiently anesthetized with local anesthetic. The tooth will be rubber dam isolated. The pulp chamber will be accessed removing all caries, defective restorations, and defective crowns. EAL and radiographs will be used to determine the working length of each canal, all canals will be cleaned and shaped using rotary files to at least a size 25.04 canal size to within 0.5 to 1 mm of the apical terminus. Between each file 5.25% NaOCl will be used to disinfect and clear the canals of debris. A final passive ultrasonic activation of NaOCl will be done for 30 seconds per canal. Each canal will then soak in 17% EDTA for 1 minute, rinsed in 5.25% NaOCl, and finally undergo a final rinse of 95% ethanol. Canals will be obturated with root canal sealer and gutta-percha.
  Arms: Standard Protocol (Control) Group

SUMMARY:
This is a clinical study that will investigate the occurrence of post-operative discomfort following the use of the Gentlewave System for root canal disinfection and irrigation. Assessment of discomfort level will be via a visualized analog pain scale.

DETAILED DESCRIPTION:
Once a tooth reaches a level of inflammation where healing can no longer occur or when the pulp space begins to go through necrosis, root canal treatment is indicated. The goal of root canal therapy is to clean, shape, disinfect, and obturate all canal systems within the tooth. Schilder's mechanical and biological objectives for cleaning and shaping includes: preparing a continuous tapering root canal funnel from access to apex, cross-sectional diameters should be wider at every point as you move coronally, the preparation should occupy as may planes as presented by the original canal and should follow the shape of the original canal, the apical foramen should remain in it is original spatial relationship to bone and to root surface, the apical opening should be kept as small as practical in all cases, complete cleaning and shaping in one appointment, procedures should be confined to the roots themselves, necrotic debris should not be forced beyond the foramina, all tissues should be removed from root canal space, and sufficient space for intracanal medicaments and irrigation should be created. Traditionally, the standard protocol for cleaning and shaping is completed using multiple hand or rotary files. Siqueira discovered that the factors that are commonly responsible for post-operative or interappointment pain include mechanical preparation and obturation beyond the apex, bacterial insults not present in the primary infection, and chemical extrusion of irrigant materials beyond the apex. Post-operative pain can occur hours to days following root canal procedures. Irrigation dissolves organic material and kills microbes. It also helps prevent the binding of instruments, improves the cutting effectiveness of files, dissolves tissue, and cools the instrument and tooth. The most common endodontic irrigant is sodium hypochlorite. Sodium hypochlorite is an alkaline fluid with a pH of approximately 11-12. It hydrolyzes proteins and causes hemolysis of red blood cells which leads to the dissolution of vital, as well as necrotic tissue. Upon contact of organic debris, hypochlorus acid forms which disrupts bacterial metabolism by oxidizing the sulfhydryl group of bacterial enzymes. The purpose of this study is to determine whether a new treatment modality for cleaning and disinfecting the root canal system will significantly affect the occurrence and severity of post-operative pain. Patients will be randomly divided into two groups, control and research. The control group will have the standard root canal procedure. The research group will have a root canal treatment that includes irrigation and disinfection with the Gentlewave system, thus eliminating the need for multiple rotatory files and multiple irrigation steps. Patients will be asked to complete a visual analog pain scale rating for pretreatment pain, as well as the same visual assessment scale for pain 6, 24, 72, & 168 hours following treatment. The results of the study should show that following Gentlewave treatment patients will experience less severe post-operative pain, if any at all. The findings should support a treatment modality that retains tooth structure while completely removing necrotic debris and bacteria, as well as causing minimal to no post-operative pain.

ELIGIBILITY:
Inclusion Criteria:

* The target population of the study includes patients needing endodontic treatment in the University of Minnesota Graduate Endodontics clinic, ages 18+. Vulnerable populations that will be included in the study are members of the military and those individuals from an undervalued or disenfranchised social group.

Exclusion Criteria:

* Patients with teeth that have root apices in the maxillary sinus, teeth with immature root apices, and teeth with insufficient coronal tooth structure will be excluded. For the purposes of this study children, pregnant women, prisoners, and adults lacking the capacity to consent will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Ordinola Zapata, DDS, MS, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, School of Dentistry Department of Graduate Endodontics, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan on sharing IPD

REFERENCES:
- [Background] Schilder H. Cleaning and shaping the root canal. Dent Clin North Am. 1974 Apr;18(2):269-96. No abstract available. PMID 4522570
- [Background] Peters OA, Peters CI, Basrani B. Cleaning and shaping the root canal system. In: Hargreaves KM, Berman LH, EDS. Cohen's pathway of the pulp. 11th ed. St. Louis: Mosby, Inc. 2016: 209-279
- [Background] Siqueira JF Jr. Microbial causes of endodontic flare-ups. Int Endod J. 2003 Jul;36(7):453-63. doi: 10.1046/j.1365-2591.2003.00671.x. PMID 12823700
- [Background] Gotler M, Bar-Gil B, Ashkenazi M. Postoperative pain after root canal treatment: a prospective cohort study. Int J Dent. 2012;2012:310467. doi: 10.1155/2012/310467. Epub 2012 Mar 15. PMID 22505897
- [Background] Haapasalo M, Shen Y, Wang Z, Gao Y. Irrigation in endodontics. Br Dent J. 2014 Mar;216(6):299-303. doi: 10.1038/sj.bdj.2014.204. PMID 24651335
- [Background] Dutner J, Mines P, Anderson A. Irrigation trends among American Association of Endodontists members: a web-based survey. J Endod. 2012 Jan;38(1):37-40. doi: 10.1016/j.joen.2011.08.013. Epub 2011 Sep 21. PMID 22152617
- [Background] Hulsmann M, Rodig T, Nordemeyer S. Complications during root canal irrigation. Endod Topics; 16: 27-63
- [Background] Pontes F, Pontes H, Adachi P, Rodini C, Almeida D, Pinto D Jr. Gingival and bone necrosis caused by accidental sodium hypochlorite injection instead of anaesthetic solution. Int Endod J. 2008 Mar;41(3):267-70. doi: 10.1111/j.1365-2591.2007.01340.x. Epub 2007 Dec 10. PMID 18081810
- [Background] Sonendo. The Gentlewave system procedure guide. 2017
- [Background] Mattscheck DJ, Law AS, Noblett WC. Retreatment versus initial root canal treatment: factors affecting posttreatment pain. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2001 Sep;92(3):321-4. doi: 10.1067/moe.2001.115135. PMID 11552152
- [Background] Menhinick KA, Gutmann JL, Regan JD, Taylor SE, Buschang PH. The efficacy of pain control following nonsurgical root canal treatment using ibuprofen or a combination of ibuprofen and acetaminophen in a randomized, double-blind, placebo-controlled study. Int Endod J. 2004 Aug;37(8):531-41. doi: 10.1111/j.1365-2591.2004.00836.x. PMID 15230906
- [Background] Sigurdsson A, Garland RW, Le KT, Rassoulian SA. Healing of Periapical Lesions after Endodontic Treatment with the GentleWave Procedure: A Prospective Multicenter Clinical Study. J Endod. 2018 Mar;44(3):510-517. doi: 10.1016/j.joen.2017.12.004. Epub 2018 Jan 12. PMID 29336878

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Protocol (Control) Group | Gentlewave Treatment Group
Started | 44 | 43
Completed | 38 | 38
Not Completed | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Protocol (Control) Group | Gentlewave Treatment Group | Total
Number analyzed (Participants) | 38 | 38 | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 28 | 56
  >=65 years | 10 | 10 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 36
  Male | 20 | 20 | 40
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Level of Post-operative Pain (2018-2019)
Description: To determine whether treatment with the Gentlewave system will significantly change the level of post-operative pain following endodontic treatment as measured by the VAS scale.
  Pain measurements were made using a 0-100 VAS- NRS. The '0' mark represented 'no pain' and the '100' mark represented 'the worst pain imaginable'. Scores 0-19 represented low pain, 20-39 was mild pain, 40-59 was moderate pain, 60-79 was high pain, and 80-100 was very high or severe pain. For this study, scores in the very high range were considered severe pain.
Time Frame: 6 hours
Measure: Mean (Standard Deviation); unit: score on VAS scale
Arm/Group | Standard Protocol (Control) Group | Gentlewave Treatment Group
Number analyzed (Participants) | 20 | 20
score on VAS scale | 23.2 (25.38) | 11.56 (9.94)

2. Primary Outcome: Level of Post-operative Pain (2018-2019)
Description: as for outcome 1
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: score on VAS scale
Arm/Group | Standard Protocol (Control) Group | Gentlewave Treatment Group
Number analyzed (Participants) | 18 | 18
score on VAS scale | 19.33 (21.46) | 7.78 (10.88)

3. Primary Outcome: Level of Post-operative Pain (2018-2019)
Description: as for outcome 1
Time Frame: 72 hours
Measure: Mean (Standard Deviation); unit: score on VAS scale
Arm/Group | Standard Protocol (Control) Group | Gentlewave Treatment Group
Number analyzed (Participants) | 18 | 18
score on VAS scale | 13.11 (18.56) | 5 (7.28)

4. Primary Outcome: Level of Post-operative Pain (2018-2019)
Description: as for outcome 1
Time Frame: 168 hours
Measure: Mean (Standard Deviation); unit: score on VAS scale
Arm/Group | Standard Protocol (Control) Group | Gentlewave Treatment Group
Number analyzed (Participants) | 18 | 18
score on VAS scale | 5.22 (10.46) | 2.78 (7.32)

5. Primary Outcome: Level of Post-operative Pain (2020-2021)
Description: as for outcome 1
Time Frame: 6 hours
Measure: Mean (95% Confidence Interval); unit: score on VAS scale
Arm/Group | Standard Protocol (Control) Group | Gentlewave Treatment Group
Number analyzed (Participants) | 20 | 20
score on VAS scale | 22 [13 to 30] | 24 [15 to 33]

6. Primary Outcome: Level of Post-operative Pain (2020-2021)
Description: as for outcome 1
Time Frame: 24 hours
Measure: Mean (95% Confidence Interval); unit: score on VAS scale
Arm/Group | Standard Protocol (Control) Group | Gentlewave Treatment Group
Number analyzed (Participants) | 20 | 20
score on VAS scale | 25 [16 to 34] | 21 [12 to 30]

7. Primary Outcome: Level of Post-operative Pain (2020-2021)
Description: as for outcome 1
Time Frame: 72 hours
Measure: Mean (95% Confidence Interval); unit: score on VAS scale
Arm/Group | Standard Protocol (Control) Group | Gentlewave Treatment Group
Number analyzed (Participants) | 20 | 20
score on VAS scale | 17 [9 to 26] | 15 [6 to 23]

8. Primary Outcome: Level of Post-operative Pain (2020-2021)
Description: as for outcome 1
Time Frame: 168 hours
Measure: Mean (95% Confidence Interval); unit: score on VAS scale
Arm/Group | Standard Protocol (Control) Group | Gentlewave Treatment Group
Number analyzed (Participants) | 20 | 20
score on VAS scale | 8 [0 to 16] | 6 [0 to 14]

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Standard Protocol (Control) Group | Gentlewave Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/38
Other Adverse Events (participants affected / at risk) | 0/38 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2018-05-07): https://cdn.clinicaltrials.gov/large-docs/15/NCT03635515/Prot_001.pdf
  • Statistical Analysis Plan (2022-10-10): https://cdn.clinicaltrials.gov/large-docs/15/NCT03635515/SAP_003.pdf
  • Informed Consent Form (2019-09-05): https://cdn.clinicaltrials.gov/large-docs/15/NCT03635515/ICF_000.pdf